CLINICAL TRIAL: NCT03116204
Title: Validation of a Score Assessing Physical and Cognitive Activities of Patients in Follow-up Care and Rehabilitation Departments: the SOFMER Activity Score
Brief Title: Validation of a SOFMER Activity Scale
Acronym: SAS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0027
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Patients Hospitalized in a FRC Department
Keywords: Dependency; FRC department; scale validation; validity; reliability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients hospitalized in a FRC department
  Interventions: Other: Assessment of score SAS

INTERVENTIONS:
Other: Assessment of score SAS — Assessment of a score assessing physical and cognitive activities of patients in follow-up care and rehabilitation departments

SUMMARY:
A person's dependency is defined as the total or partial inability to perform without helps the necessary activities of daily life due to activity limitations in the usual environment. The consequence is a restriction of participation. In physical and Rehabilitation Medicine (PRM), dependency impacts the healthcare team activity at several levels: patient's referral and care plan, conditions of home return and resumption of course of life, burden of care assessment and care teams management...

The main goal of this project is the validation of a score assessing physical and cognitive activities of patients in follow-up care and rehabilitation (FRC) departments based on the ICF model (International Classification of Functioning, Disability and Health) : the SOFMER Activity Scale (SAS).

We want to propose a French generic scale allowing quantifying precisely the dependence and burden of care of patients in FRC departments. This scale needs to be valid, easy to apply, easy to learn, reproducible, sensitive to change and common to adult subjects, children and elderly.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 2 years old
* Hospitalized in the participating department for at least 4 days
* For the responsiveness study : patients hospitalized in the FRC departments for obesity, spinal cord injuries, post-stroke rehabilitation or cardiorespiratory rehabilitation after cardiac surgery

Exclusion Criteria:

* Non-recipient of French Social Security

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in a FRC department
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Assessment of the validity of SAS | Day 0
  The construct validity will be determined by an exploratory factor analysis and confirmed on an independent sample.
  Criterion validity will be studied by comparison of scores obtained from SAS to scores obtained from references scale (FIM, WeeFIM, ADL, IADL, BREF, BREV, MMSE and items of WISC IV).
Assessment of the reliability of SAS. | Day 7
  For the inter rater reliability study, patients will be rated on the same day by two groups of therapists.
  For the test-retest reliability study, patients will be rated twice during their hospitalization, within a time frame sufficiently close so that their dependency should not change.

SECONDARY OUTCOMES:
Study of SAS responsiveness | 6 months
  Sensitivity to change will be studied on patients hospitalized in a FRC departments for obesity, spinal cord injuries, post-stroke rehabilitation or cardiorespiratory rehabilitation after cardiac surgery. The change between scores of SAS at entry and exit (or at maximum 6 months after inclusion) of hospitalization will be studied.
Study of invariance of SAS: invariance of the classification between age and sex classes. | day 0
  Invariance of SAS will be determined between three age classes (<18 years, 18-75 years,> 75 years) using three confirmatory factor analyzes

CONTACTS AND LOCATIONS:
Overall Officials: Carole VUILLEROT, Principal Investigator — Hospices Civils de Lyon
Locations (9):
- France (9):
  - Centre SSR Les Capucins, Angers
  - Etablissement Hopale-Centre Calvé, Berck
  - Service SSRS Enfants et Adolescents, Fondation Ildys, Brest
  - Département de Rééducation Neurologique - Hôpital Sud - CHU de Grenoble, Échirolles
  - Médecine physique et réadaptation - Hôpital Raymond Poincaré - APHP, Garche
  - Ctre Médico-Chir Réadapt Des Massues, Lyon
  - Service de Médecine physique et Réadaptation - Hôpital Henry Gabrielle, Lyon
  - Service de Médecine Physique et de Réadaptation - F.Widal - APHP, Paris
  - Service de Médecine Physique et Réadaptation - Pôle Couple Mère-Enfant - HOPITAL DE BELLEVUE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No